CLINICAL TRIAL: NCT03747172
Title: Use of Complementary and Alternative Medicine by Hospice Oncology Patients During Ambulatory Palliative Care
Brief Title: Use of CAM by Hospice Oncology Patients During Ambulatory Palliative Care
Acronym: CAM
Status: Completed | Type: Observational
Sponsor: Silesian University of Medicine (Other)
Responsible Party: Principal Investigator, Łukasz Pietrzyński, Principal Investigator, Silesian University of Medicine
Other Study IDs: CAM001
Record Dates: First submitted 2018-10-23; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Complementary Alternative Medicine; Complementary Alternative Therapy; Hospice Care
Keywords: complementary alternative medicine; cancer; complementary alternative therapy; hospice care; palliative care
MeSH Terms: conditions — Neoplasms | interventions — Complementary Therapies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: complementary and alternative therapy — complementary and alternative therapies were grouped into five main categories: (1) biologically based therapies , (2) mind/body therapies, (3) manipulative and body-based therapies, (4) Energy therapies and (5) alternative medical systems.

SUMMARY:
The aim of the study is to assess Prevalence of complementary and alternative therapy use by adult patients from the area of Silesian agglomeration (Poland) with advanced, metastatic cancer disease who were admitted to "Pro Salute" Hospice for ambulatory palliative care between July 2017 and September 2018

DETAILED DESCRIPTION:
The research team developed the CAT (complementary and alternative therapy) screening tool to obtain information about CAM use from patients. The screening tool was based on a The National Center for Complementary and Alternative Medicine's (NCCAM) classification of CAM. CAT were grouped into five main categories: (1) biologically based therapies , (2) mind/body therapies, (3) manipulative and body-based therapies, (4) Energy therapies and (5) alternative medical systems.

The questionaire was tailored to meet the objectives of this study and to be adjusted to hospice patients specifics. It was piloted on the group of 25 patients, resulting in some vocabulary changes. The final questionnaire consists of 25 multiple-choice, semi-structured questions and takes about 15 min to complete. For each general CAM category the detailed information was collected on the type of specific therapy that was used. Patients were considered as CAM users if they have used at least one therapy from at least one of the categories during the period of 12 months prior to the screening. Patients were asked to specify the reasons for CAT usage, experienced effects of the therapy, stage at which patients considered using CAM

ELIGIBILITY:
Inclusion Criteria:

* adult patients from the area of Silesian agglomeration (Poland) with advanced, metastatic cancer disease who were admitted to "Pro Salute" Hospice for ambulatory palliative care between July 2017 and September 2018

Exclusion Criteria:

* Patients were excluded from the survey if they presented cognitive disturbances disabling credible answers in the questionnaire

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients from the area of Silesian agglomeration (Poland) with advanced, metastatic cancer disease who were admitted to "Pro Salute" Hospice for ambulatory palliative care between July 2017 and September 2018
Sampling Method: Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Variation of prevalence of complementary and alternative therapy use by hospice patients | 14 months
  Presence and quantity of patients using any CAM therapies -The research team developed the CAT screening tool based on a The National Center for Complementary and Alternative Medicine's (NCCAM) classification of CAM. Questionnaire consists of 25 multiple-choice, semi-structured questions and gives the result in the form of a percentage
Variation of prevalence of biologically based therapies | 14 months
  Presence and quantity of patients using biologically based therapies - The research team developed the CAT screening tool based on a The National Center for Complementary and Alternative Medicine's (NCCAM) classification of CAM. Questionnaire consists of 25 multiple-choice, semi-structured questions and gives the result in the form of a percentage
Variation of prevalence of mind/body therapies | 14 months
  Presence and quantity of patients using mind/body therapies - The research team developed the CAT screening tool based on a The National Center for Complementary and Alternative Medicine's (NCCAM) classification of CAM. Questionnaire consists of 25 multiple-choice, semi-structured questions and gives the result in the form of a percentage
Variation of prevalence of manipulative and body-based therapies | 14 months
  Presence and quantity of patients using manipulative and body-based therapies - The research team developed the CAT screening tool based on a The National Center for Complementary and Alternative Medicine's (NCCAM) classification of CAM. Questionnaire consists of 25 multiple-choice, semi-structured questions and gives the result in the form of a percentage
Variation of prevalence of biologically Energy therapies | 14 months
  Presence and quantity of patients using Energy therapies - The research team developed the CAT screening tool based on a The National Center for Complementary and Alternative Medicine's (NCCAM) classification of CAM. Questionnaire consists of 25 multiple-choice, semi-structured questions and gives the result in the form of a percentage
Variation of prevalence of alternative medical systems | 14 months
  Presence and quantity of patients using alternative medical systems - The research team developed the CAT screening tool based on a The National Center for Complementary and Alternative Medicine's (NCCAM) classification of CAM. Questionnaire consists of 25 multiple-choice, semi-structured questions and gives the result in the form of a percentage

CONTACTS AND LOCATIONS:
Locations (1):
- PZZOZ Będzin, Będzin, Poland

IPD SHARING:
Plan to Share IPD: No